CLINICAL TRIAL: NCT05760586
Title: Expanded Access to the Oral Pan-RAF Inhibitor DAY101 in Pediatric Patients With RAF-Altered, Relapsed or Refractory Low-Grade Glioma
Brief Title: Expanded Access Program (EAP) for Tovorafenib (DAY101) in RAF-Altered, Relapsed or Refractory Low-Grade Glioma
Status: Approved for marketing | Type: Expanded Access
Sponsor: Day One Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DAY101-EAP
Record Dates: First submitted 2023-02-02; First posted 2023-03-08 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Low-grade Glioma
Keywords: DAY101; Toverafenib; Glioma; BRAF Mutation; RAF Alteration; Type II BRAF Inhibitor; Neoplasms
MeSH Terms: conditions — Glioma; Neoplasms | interventions — tovorafenib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Tovorafenib — Oral RAF inhibitor provided as an immediate-release tablet (100 mg) or powder for reconstitution (25 mg/mL)
  Other Names: DAY101

SUMMARY:
The DAY101-EAP is a multicenter, open-label, expanded access treatment protocol designed to provide access to tovorafenib (DAY101) for eligible patients.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for enrollment in the EAP:

1. Patients must be aged 6 months to 25 years, inclusive, with a relapsed or refractory low-grade glioma with a documented known or expected to be activating BRAF mutation or RAF fusion, as identified through molecular assays as routinely performed at CLIA-certified or other similarly certified laboratories.
2. Patients must have histopathologic diagnosis of glioma or glioneuronal tumor (Grade 1 or 2 according to WHO classification for CNS tumors at either original diagnosis or relapse.
3. Patients must have received at least one line of prior systemic therapy and have documented evidence of radiographic progression.
4. Previous chemotherapy and/or targeted/immunotherapy/monoclonal antibody therapy must be completed at least 4 weeks or 5 half-lives (whichever is shorter) prior to the initiation of therapy.
5. Chronic toxicities from prior anticancer therapy must be stable and at CTCAE Version 5.0 Grade ≤ 2.
6. Patients must have fully recovered from any prior surgery.
7. Patients must have adequate hematologic function, as defined by the following:

   1. Absolute neutrophil count≥ 1000/mm3
   2. Platelet count≥ 75.0 × 109/L
   3. Hemoglobin≥ 10.0 g/dL (transfusions allowed up to 14 days prior to enrollment per institutional guidelines)
8. Patients must have adequate hepatic and renal function, defined by the following:

   1. Total bilirubin ≤ 1.5 × upper limit of normal (ULN) for age (If patient has documented Gilbert's Disease, patient may be enrolled with Sponsor approval, provided that bilirubin is < 2.0 × ULN)
   2. Serum glutamic-pyruvic transaminase (SGPT)/alanine aminotransferase (ALT) ≤ 3 × ULN
   3. Serum glutamic-oxaloacetic transaminase (SGOT)/aspartate transaminase (AST) ≤ 3 × ULN
   4. Serum creatinine within normal limits, or estimated glomerular filtration rate ≥ 60 mL/min/1.73 m2 based on local institutional practice for determination
9. Thyroid function tests must be consistent with stable thyroid function.
10. Patients must be able to comply with treatment, laboratory monitoring, and required clinic visits for the duration of EAP participation.
11. Male and female patients with reproductive potential must be willing to use birth control methods per Appendix E of protocol.
12. Patients must be able to swallow tablets or liquid or administer through gastric access via feeding tube(12Fr or greater)
13. Parent/guardian of child or adolescent patient must have the ability to understand, agree to, and sign the EAP informed consent form (ICF) and applicable pediatric assent form before initiation of any treatment-related procedures; patient must have the ability to give assent, as applicable, at the time of parental/guardian consent.

Exclusion Criteria:

Patients meeting any of the following criteria are to be excluded from EAP participation:

1. Patient's tumor has an additional previously known or expected to be activating molecular alteration(s) (e.g., histone mutation, IDH1/2 mutations, FGFR mutations or fusions, MYBL alterations, neurofribromatosis type 1 (NF-1) somatic or germline mutations).
2. Patient has known or suspected diagnosis of neurofibromatosis type 1 (NF-1) via genetic testing or current diagnostic criteria.
3. Patient has history of any major disease, other than the primary malignancy under EAP, that might interfere with safe protocol participation.
4. Patient has major surgery within 14 days (2 weeks) prior to C1D1 (does not include central venous access, cyst fenestration or cyst drainage, or ventriculoperitoneal shunt placement or revision).
5. Patient has clinically significant active cardiovascular disease, or history of myocardial infarction, or deep vein thrombosis/pulmonary embolism within 6 months prior to C1D1, ongoing cardiomyopathy, or current prolonged QT interval corrected for heart rate by Fridericia's formula (QTcF) interval > 470 milliseconds based on triplicate electrocardiogram (ECG) average.
6. Patient has an active systemic bacterial, viral, or fungal infection.
7. Patient has malabsorption requiring supplementation, or significant bowel or stomach resection that would preclude adequate absorption of tovorafenib (DAY101).
8. Concomitant medications that are strong inhibitors or inducers of CYP2C8 within 14 days before initiation of therapy. Concomitant medications that are substrates of BCRP with a narrow therapeutic index within 14 days before initiation of therapy.
9. Patient is pregnant or lactating, or plans to become pregnant in the immediate future.
10. Patient has any clinically significant skin toxicity at screening, that in the opinion of the investigator would increase risk of severe skin toxicity when using investigational product.
11. There are other unspecified reasons that, in the opinion of the HCP, make the patient unsuitable for enrollment.
12. Patient has CTCAE v5.0 Grade ≥3, CPK elevation ( > 5x UL - 10 X ULN)

Ages: 6 Months to 25 Years | Sex: All
Age Groups: Child, Adult